CLINICAL TRIAL: NCT04717323
Title: Precision Gait Retraining for Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altec Inc. (Industry)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: mPAD Phase 1
Record Dates: First submitted 2020-12-07; First posted 2021-01-22 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Cerebral Palsy; Gait Disorders, Neurologic
Keywords: CP (Cerebral Palsy); Diplegia, Spastic; Gait Disorders
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): Gait with and without pelvic assistance
  Interventions: Device: mPAD (or TPAD) Pelvic Assist Device; Device: No Intervention
- Controls (Experimental): Gait with no pelvic assistance
  Interventions: Device: No Intervention

INTERVENTIONS:
Device: mPAD (or TPAD) Pelvic Assist Device — Gait retraining device that applies pelvic forces and measures response
  Other Names: mPAD (or TPAD)
  Arms: Patients
Device: No Intervention — Gait with no pelvic assistance

SUMMARY:
This project will develop the first sensor-based mobile Pelvic Assist Device (mPAD) that can deliver precise, adaptable, pelvic control to restore natural coordination of upper- and lower-limb movements during gait in children with Cerebral Palsy

DETAILED DESCRIPTION:
Gait impairments hinder mobility for more than 760,000 children and adults living with cerebral palsy (CP) in the US. Motor relearning is possible for these individual but typically requires numerous training sessions with a team of physical therapists and assistants to restore coupling between upper- and lower-body segments while assisting spastic uncoordinated limb movement to improve gait kinematics. This clinical trial will meet the overall objective of testing the feasibility of developing a smart-robotic exoskeleton that is effective at providing guided pelvic assistance and support while biofeedback mediated training is facilitated under the supervision of a physiotherapist. The project will test a novel tethered Pelvic Assist Device (TPAD) with integratable electromyographic (EMG) and inertial (IMU) biofeedback that is uniquely capable of delivering precise, adaptable, multi-degree-of-freedom pelvic control to promote natural intersegmental coupling, restore coordination of upper- and lower-limb movement, and improve normal gait kinematics in children with CP. Because of its proximity to the center of mass and critical role in coordinating upper- and lower-limb control, the pelvis provides an ideal access point for physiotherapists to manually improve gait. The investigators will test the hypothesis that accurate sensor-based metrics of gait can be derived from EMG and IMU wearable sensors to develop a biofeedback system for motor learning that are integratable with TPAD to develop a new mobile mPAD device that is compliant with the target population.

ELIGIBILITY:
Inclusion Criteria (children with CP):

* Children (6-18 years of age)
* Male or Female
* Confirmed diagnosis of Cerebral Palsy by a neurologist;
* CT or MRI imaging consistent with clinical presentation;
* Clinical evidence of preserved cognition as determined by the child's neurologist;
* Clinical evidence of Mild to Moderate spastic (pyramidal) diplegia as determined by the child's neurologist;
* Gross Motor Function Classification System (GMFS) GMFCS Level II ("walks with limitations. Limitations include walking long distances and balancing, but not as able as Level I to run or jump; may require use of mobility devices when first learning to walk, usually prior to age 4; and may rely on wheeled mobility equipment when outside of home for traveling long distances."
* Spasticity being controlled by pharmaceutical or surgical correction; or has Modified Ashworth scale (MAS) = 0-2 ("More marked increase in muscle tone through most of the range of motion (ROM), but affected part(s) easily moved
* Ambulatory without assistive devices (except for long distances or on uneven terrain).
* No allergies to skin tape such as Band-Aid.

Exclusion Criteria (children with CP):

* Inability to follow simple instructions in English, or through a Spanish-speaking translator;
* Medical history of other neurological conditions;
* Medical history of cardiac or respiratory complications, or disorders that would place the subject at risk for conducting the different motor activities;
* Contractures present in lower limb - evaluated based on Tardieu Scale test where joint range of motion is measured during slow velocity movements and where contracture is operationally defined as being present if the angle at the end of range is 5 -10 degrees less than full range at ankle; and 5 -20 degrees less than full range at hip and knee.
* Skin disorders that result in open lesions or hyper-sensitive/fragile skin, preventing the use of medical-grade adhesive tapes to secure the sensors to the skin;
* Unable to provide Informed Consent from subject and Assent from parent or guardian using English or Spanish-translation informed consent form.

Inclusion Criteria (healthy volunteers):

* Adults or Children (age≥6 y.o.)
* Male or Female;
* Able to walk independently and without assistive devices;
* No history of musculoskeletal or neurological disorders;
* Able to follow directions in English.

Exclusion criteria (healthy volunteers):

* Non-English speaker;
* Unable to walk independently and without assistive devices;
* Medical history of neurological or musculoskeletal conditions (arthritis, spondylosis, etc.);
* Inability to follow simple instructions;
* Unable to provide informed consent in English.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Contessa, PhD, Principal Investigator — Altec Inc.
Locations (2):
- United States (2):
  - Altec Inc., Natick, Massachusetts
  - CUMC Harkness Pavillion, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be made through conferencing

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients | Controls
Started | 0 | 10
Completed | 0 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes only controls that participated in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients | Controls | Total
Number analyzed (Participants) | 0 | 10 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 10 | 10
  >=65 years |  | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 27.3 (2.8) | 27.3 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 5 | 5
  Male |  | 5 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 10 | 10
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 2 | 2
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 8 | 8
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 10 | 10

OUTCOME MEASURES:

1. Primary Outcome: Gait Metric Accuracy
Description: Measures the accuracy of identifying heel strike and toe off timing in % error when comparing measures from wearable sensors vs. motion capture
Time Frame: 1 day
Population: Analysis was conducted for control participants that completed the study procedure.
Measure: Mean (Standard Deviation); unit: percentage of error
Arm/Group | Patients | Controls
Number analyzed (Participants) | 0 | 10
percentage of error |  | 2.01 (1.44)

2. Primary Outcome: Pelvis Range of Motion During Walking
Description: Difference (in degrees) between pelvis range of motion during walking as detected by wearable sensors and motion capture
Time Frame: 1 day
Population: Analysis was conducted for control participants that completed the study procedure
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Patients | Controls
Number analyzed (Participants) | 0 | 10
degrees |  | 1.40 (0.60)

3. Primary Outcome: Muscle Activation During Walking
Description: Measures electromyographic (EMG) signals of trunk and lower limb muscles during gait which are necessary for designing and implementing a mobile pelvic assist device (mPAD) system with biofeedback
Time Frame: 1 day
Population: Analysis was not conducted since patient participants in need of EMG biofeedback were not recruited.
Arm/Group | Patients | Controls
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Rating of Perceived Difficulty
Description: Structured interviews will be used to grade the perception of difficulty in using the technology
Time Frame: 1 day
Population: Analysis was not conducted since patient participants assigned to the pelvic assistance intervention were not recruited.
Arm/Group | Patients | Controls
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Trunk Range of Motion During Walking
Description: Difference (in degrees) between trunk range of motion during walking as detected by wearable sensors and motion capture
Time Frame: 1 day
Population: Analysis was conducted for control participants that completed the study procedure
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Patients | Controls
Number analyzed (Participants) | 0 | 10
degrees |  | 1.34 (0.50)

6. Primary Outcome: Hip Range of Motion During Walking
Description: Difference (in degrees) between hip range of motion during walking as detected by wearable sensors and motion capture
Time Frame: 1 day
Population: Analysis was conducted for control participants that completed the study procedure
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Patients | Controls
Number analyzed (Participants) | 0 | 10
degrees |  | 2.09 (0.90)

7. Primary Outcome: Knee Range of Motion During Walking
Description: Difference (in degrees) between knee range of motion during walking as detected by wearable sensors and motion capture
Time Frame: 1 day
Population: Analysis was conducted for control participants that completed the study procedure
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Patients | Controls
Number analyzed (Participants) | 0 | 10
degrees |  | 3.12 (1.27)

ADVERSE EVENTS:
Time Frame: Through assessment duration, an average of 1 day
Description: Includes only controls that participated in the study.
Groups:
- Pelvic Assist (Patients): Pelvic assistance applied for gait retraining
  mPAD (or TPAD) Pelvic Assist Device: Gait retraining device that applies pelvic forces and measures response
  No Intervention: Gait with no pelvic assistance
- No Intervention (Controls): Gait with no pelvic assistance
  No Intervention: Gait with no pelvic assistance
Arm/Group | Pelvic Assist (Patients) | No Intervention (Controls)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/10
Other Adverse Events (participants affected / at risk) | 0/0 | 0/10

LIMITATIONS AND CAVEATS:
Intervention was not assigned due to mandated patient recruitment restrictions resulting from the Covid-19 emergency.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT04717323/Prot_SAP_000.pdf